CLINICAL TRIAL: NCT06075030
Title: A Multicenter, Randomized, Open-label Study of AND017 for the Treatment of Cancer-Related Anemia Patients Receiving Chemotherapy
Brief Title: A Study of AND017 in Cancer Related Anemic Patients Receiving Chemotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kind Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AND017-CRA-201
Record Dates: First submitted 2023-03-22; First posted 2023-10-10 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Chemotherapy Induced Anemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AND017 Dose A three times weekly (Experimental)
  Interventions: Drug: AND017
- AND017 Dose B three times weekly (Experimental)
  Interventions: Drug: AND017
- AND017 Dose C three times weekly (Experimental)
  Interventions: Drug: AND017

INTERVENTIONS:
Drug: AND017 — Oral administration of AND017 capsules three times per week

SUMMARY:
The purpose of this study is to determine the safety and efficacy of AND017 after 6 weeks of treatment in patients with cancer-related anemia who are receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Non-myeloid malignancy diagnosed by cytology/histology
2. Receiving and have received at least one cycle of drug therapy with a high myelosuppressive adverse effect, including but not limited to chemotherapeutic agents such as platinum, targeted agents, antibody-coupled drugs, immunosuppressive agents, etc., and are expected to continue such therapy within 8 weeks of enrollment
3. ECOG score of 0-2 and an expected survival of 6 months or more.
4. Mean hemoglobin <10.0 g/dL at screening test and one follow-up test (at least one week thereafter during the screening period), with a difference between the two tests of ≤1.0 g/dL
5. Total bilirubin <1.5 x upper limit of normal (ULN) If Gilbert's syndrome (unconjugated hyperbilirubinemia) have a total bilirubin < 3 x ULN.
6. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x ULN.
7. No iron deficiency, TSAT ≥ 20% and ferritin ≥ 100 ng/mL at screening.
8. Serum folate and vitamin B12 ≥ lower limit of normal at screening.
9. eGFR >60 mL/min/1.73 at screening.

Exclusion Criteria:

1. Hematocrit (Hct) ≥ 36 vol% at the screening assessment.
2. Prior history of leukemia.
3. Extensive bone metastases from breast cancer, head and neck cancer with combined whole blood (trilineage) cytopenia, bone marrow invasion from lymphoma, definite brain metastases (except for those whose symptoms have been controlled for ≥4 weeks) or bone marrow metastases.
4. Combination of hereditary anemia, iron-granulocytic anemia, acute blood loss, active bleeding (three consecutive positive fecal occult bloods or clinical judgment of the investigator), hemolysis and other diseases that can cause anemia such as iron, folic acid or vitamin B12 deficiency.
5. Active infection or inflammatory disease requiring systemic anti-infective therapy within 1 week prior to the first dose, including concurrent autoimmune diseases with inflammatory symptoms (e.g., generalized erythema, ankylosing spondylitis, rheumatoid arthritis, psoriatic arthritis, dry syndrome, celiac disease, etc.)
6. Concurrent retinal neovascularization requiring treatment (diabetic proliferative retinopathy, age-related exudative macular degeneration, retinal vein occlusion, macular edema, etc.)
7. Difficulty to take oral medications, or conditions that may have an impact on the absorption of gastrointestinal medications such as a history of gastrectomy/bowel resection or concomitant gastroparesis (excluding gastric polyps or colonic polypectomy).
8. clinically significant bleeding (including the need for blood transfusion or a decrease in hemoglobin ≥ 2 g/dL) within 4 weeks prior to the first dose, or a bleeding constitutional or bleeding risk that has not been medically or surgically corrected.
9. Uncontrolled hypertension (more than one-third of identifiable diastolic blood pressure values > 90 mmHg and/or systolic blood pressure ≥ 160 mmHg at 16 weeks prior to and including screening testing)
10. Concurrent congestive heart failure (New York Heart Association [NYHA] class III or higher).
11. Clinically significant ECG abnormalities at the time of screening evaluation
12. Medical history of significant liver disease or active liver disease
13. History of stroke, transient ischemic attack (TIA), myocardial infarction, thromboembolic event (deep vein thrombosis, DVT), pulmonary embolism, or pulmonary infarction within 24 weeks prior to the screening evaluation
14. History of prior thrombosis, significant coagulation abnormalities, history of hematologic disease, or history of ineffective erythropoietin therapy
15. History of epilepsy or any past seizures.
16. Positive hepatitis B surface antigen (HBsAg), or positive anti-hepatitis C virus (HCV) antibodies, or positive human immunodeficiency virus HIV at screening evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of responding patient | From baseline to Week 6 or End of Treatment visit
  Responding patient is defined as those with a maximum change from baseline in hemoglobin level greater than 10% during the treatment

SECONDARY OUTCOMES:
Transfusion treatment rate | From baseline to Week 6 or End of Treatment visit
  The percentage of subjects who need to receive blood transfusion during the treatment
Mean and change from baseline in hemoglobin levels at each study visit | From baseline to Week 6 or End of Treatment visit
  Mean and change from baseline in hemoglobin levels at each study visit
The maximum change from baseline in hemoglobin during the treatment | From baseline to Week 6 or End of Treatment visit
  The maximum change from baseline in hemoglobin during the treatment
Percentage of visits in which subjects maintained a hemoglobin between elevation >10% of baseline and hemoglobin<12.0 g/dL after reaching an elevation of 10% from baseline | From baseline to Week 6 or End of Treatment visit
  Percentage of visits in which subjects maintained a hemoglobin between elevation >10% of baseline and hemoglobin<12.0 g/dL after reaching an elevation of 10% from baseline
Percentage of subjects whose hemoglobin remained between elevation >10% of baseline and hemoglobin< 12.0 g/dL after 5 weeks treatment | At baseline and Week 6
  Percentage of subjects whose hemoglobin remained between elevation >10% of baseline and hemoglobin< 12.0 g/dL after 5 weeks treatment
Time for hemoglobin reaching an elevation of >10% from baseline during treatment | From baseline to Week 6 or End of Treatment visit
  Time for hemoglobin reaching an elevation of >10% from baseline during treatment